CLINICAL TRIAL: NCT05897684
Title: Avacostar - A Post Authorization Safety Study (PASS) to Evaluate the Incidence of Safety Events of Interest in Patients Treated With Avacopan for ANCA-associated Vasculitis (AAV)
Brief Title: Avacostar - (PASS)
Acronym: Avacostar
Status: Recruiting | Type: Observational
Sponsor: Vifor Fresenius Medical Care Renal Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-AVA-2022-0016
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: ANCA-associated Vasculitis
Keywords: anti-neutrophil cytoplasmic antibody (ANCA)-AAV
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: US Export: Yes

GROUPS / COHORTS (2):
- Treated with avacopan for active AAV: The study will enrol approximately 250 adult patients diagnosed with AAV (MPA or GPA) treated with avacopan for active severe AAV.
- Treated with a cyclophosphamide or rituximab-based induction regimen without avacopan for active AAV: The study will enrol approximately 250 adult patients diagnosed with AAV (MPA or GPA) treated with a cyclophosphamide or rituximab-based induction regimen without avacopan for active severe AAV.

SUMMARY:
The Avacostar PASS is a non-interventional, multi-national, prospective cohort study that will collect data from 2 cohorts of patients: those treated with avacopan for active severe AAV, and a second cohort treated with a cyclophosphamide or rituximab-based induction regimen without avacopan for active severe AAV. The overall study duration is anticipated to be up to 7 years, including a recruitment period of approximately 3 years.

DETAILED DESCRIPTION:
The Avacostar PASS is a non-interventional, multi-national, prospective cohort study that will collect data from 2 cohorts of patients: those treated with avacopan for active severe AAV, and a second cohort treated with a cyclophosphamide or rituximab-based induction regimen without avacopan for active severe AAV. The overall study duration is anticipated to be up to 7 years, including a recruitment period of approximately 3 years. Enrolled patients will be followed until the last patient last visit (LPLV) milestone, which will be 4 years after the last participant is enrolled.

Germany and the United Kingdom (UK) have been selected for the study. Additional countries may be considered according to availability of avacopan and suitability for the study. Patients will be enrolled prospectively, but up to 6 months of data may be collected retrospectively if necessary. Baseline visit is defined as the day that induction treatment (avacopan or non-avacopan standard of care (SoC) cyclophosphamide or rituximab) is started for active severe AAV. Patients who started avacopan/SoC induction therapy for active severe AAV within 6 months of the enrolment visit and fulfil eligibility criteria may be enrolled in the PASS. Individual participant follow-up data will be collected periodically at routine clinic visits until the LPLV, which will be 4 years after the last participant is enrolled.

The primary objective of the study is:

To evaluate the incidence of defined Medical Events of Special Interest (MESIs) in patients with AAV commencing avacopan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AAV (MPA or GPA), as determined by the Investigator according to their usual practice.
* Active, severe AAV at the time of commencing avacopan or non-avacopan SoC induction therapy, in the opinion of the Investigator.
* Age ≥18 years of either sex.
* Has provided written informed consent.
* Has commenced within the previous 6 months, or is planned to commence avacopan, cyclophosphamide or rituximab for the treatment of severe, active AAV outside of an interventional clinical study.

Exclusion Criteria:

• Concurrent participation in an interventional study, unless prospectively discussed and agreed with the Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Avacostar PASS is a non-interventional, multi-national, prospective cohort study that will collect data from 2 cohorts of patients: those treated with avacopan for active severe AAV, and a second cohort treated with a cyclophosphamide or rituximab-based induction regimen without avacopan for active severe AAV.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence of defined MESIs | up to 7 years
  To evaluate the incidence of defined MESIs in patients with AAV commencing avacopan. MESIs include liver injury, cardiac safety, serious infection, and malignancy.

SECONDARY OUTCOMES:
Incidence rates of AE in the avacopan and non-avacopan groups | up to 7 years
AEs leading to discontinuation of therapy in the avacopan group | up to 7 years
Incidence of SAEs in the avacopan and non-avacopan groups | up to 7 years
Incidence of ADRs in the avacopan group | up to 7 years
Incidence of SADRs in the avacopan group | up to 7 years
Change in eGFR over time in the avacopan and non-avacopan groups | up to 7 years
Change in IgG over time in the avacopan and non-avacopan groups | up to 7 years
Change in CPK over time in the avacopan and non-avacopan groups | up to 7 years
Change in ALT over time in the avacopan and non-avacopan groups | up to 7 years
Change in AST over time in the avacopan and non-avacopan groups | up to 7 years
Change in billirubin over time in the avacopan and non-avacopan groups | up to 7 years
Change in WBC over time in the avacopan and non-avacopan groups | up to 7 years
Change Albumin over time in the avacopan and non-avacopan groups | up to 7 years
Time to first flare over time in the avacopan and non-avacopan groups | up to 7 years
  A flare is defined in the BVAS as a score of more than 0. No flare is defined as a BVAS score equal to 0
Change in VDI scores over time in the avacopan and non-avacopan groups | up to 7 years
Incidence of MESIs in the non-avacopan group | up to 7 years
Incidence rates of SAEs and MESIs in the avacopan group compared to the non-avacopan group, | up to 7 years
Incidence rates of MESIs in the avacopan group compared to the non-avacopan group, | up to 7 years
Use of concomitant immunosuppression over time and cumulative by treatment group, | up to 7 years
Duration of GC-free periods | up to 7 years
Proportion of GC-free patients over time by treatment group. | up to 7 years
Duration of treatment with avacopan by reason for treatment discontinuation. | up to 7 years

CONTACTS AND LOCATIONS:
Locations (35):
- Germany (12):
  - Charité University Medicine, Berlin
  - University Hospital of Cologne, Cologne
  - Municipal Hospital Dresden, Dresden
  - University Hospital Essen, Essen
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Medical Center Göttingen, Göttingen
  - University Hospital Eppendorf, Hamburg
  - KRH Klinikum Siloah, Hanover
  - Rheumazentrum Ruhrgebiet, Herne
  - LMU, Munich
  - Medius Kliniken, Plochingen
  - St. Josef-Stift Sendenhorst, Sendenhorst
- United Kingdom (23):
  - UHB NHS Foundation Trust, Birmingham
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - North Bristol NHS Trust, Bristol
  - Addenbrookes Hospital, Cambridge
  - East Kent Hospitals University NHS FT, Canterbury
  - Cardiff and Vale UHB, Cardiff
  - Epsom & St. Helier NHS Trust, Carshalton
  - University Hospitals Coventry and Warwickshire, Coventry
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - NHS Greater Glasgow & Clyde, Glasgow
  - University Hospitals of Leicester NHS Trust, Leicester
  - Barts Health, London
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London
  - Kings College Hospital, London
  - Royal Free, London
  - St Thomas' Hospital, London
  - Manchester University NHS Foundation Trust, Manchester
  - Nottingham university hospitals NHS trust, Nottingham
  - Rheumatology Department, Oxford University Hospitals NHS Foundation Trust, Oxford
  - Royal Berkshire NHS foundation trust, Reading
  - Northern Care Alliance, Salford
  - Swansea Bay University LHB, Swansea
  - York & Scarborough Teaching Hospitals NHS FT, York

IPD SHARING:
Plan to Share IPD: No